CLINICAL TRIAL: NCT05659420
Title: The Effect of High-intensity Interval Training and Moderate Intensity Continuous Training on Cardiopulmonary Functions in Chronic Heart Failure
Brief Title: High Intensity Interval Training in Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Joa KyungLim, professor, M.D. Ph.D, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: InhaUH
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Chronic Heart Failure; Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity interval training (Experimental)
  Interventions: Behavioral: Cardiac rehabilitation comprised aerobic exercise on a treadmill accompanied by an electrocardiogram monitoring device and a blood pressure monitor
- Moderate intensity continous training (Active Comparator)
  Interventions: Behavioral: Cardiac rehabilitation comprised aerobic exercise on a treadmill accompanied by an electrocardiogram monitoring device and a blood pressure monitor
- Control (Placebo Comparator)
  Interventions: Behavioral: Cardiac rehabilitation comprised aerobic exercise on a treadmill accompanied by an electrocardiogram monitoring device and a blood pressure monitor

INTERVENTIONS:
Behavioral: Cardiac rehabilitation comprised aerobic exercise on a treadmill accompanied by an electrocardiogram monitoring device and a blood pressure monitor — aerobic exercise on a treadmill (T7M, Motus, Paju, South Korea) accompanied by an electrocardiogram monitoring device (Q-Tel Rehabilitation Management System, Mortara Inc., Milwaukee, WI, USA) and a blood pressure monitor

SUMMARY:
The aim of this study is to investigate the effect of high-intensity interval training and moderate intensity continuous training on cardiopulmonary functions in chronic heart failure.

DETAILED DESCRIPTION:
enroll chronic heart failure patients into 3 randomized controlled group

* high intensity interval training
* moderate intensity continous training
* control

perform cardica rehab for 12 weeks, compare primary and secondary endpoints between baseline and 12 weeks results

ELIGIBILITY:
Inclusion Criteria:

* medically stable chronic heart failure
* NYHA II-III
* can perform cardiopulmonary exercise test
* after 3months with proper medication
* age 30 to 70
* ejection fraction< 40%

Exclusion Criteria:

* contraindication to cardiopulmonary exercise test
* musculoskeletal problem who cannot perform cardiopulmonary exercise test
* cognition deficit who cannot understand directions
* severe medial illness

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal or peak oxygen consumption (VO2max or VO2peak, same meaning) (kg/ml/min) | compare baseline data with 12 weeks rehabilitation data
  at the end of training, from baseline to 12 weeks

SECONDARY OUTCOMES:
Anaerobic threshold (kg/ml/min) | compare baseline data with 12 weeks rehabilitation data
  The anaerobic threshold is the highest exercise intensity that you can sustain for a prolonged period without lactate substantially building up in your blood.
6minute walk test (meter) | compare baseline data with 12 weeks rehabilitation data
maximal heart rate (bpm) | compare baseline data with 12 weeks rehabilitation data
systolic blood pressure (mmHg) | compare baseline data with 12 weeks rehabilitation data
diastolic blood pressure (mmHg) | compare baseline data with 12 weeks rehabilitation data
resting heart rate (bpm) | compare baseline data with 12 weeks rehabilitation data
diastolic blood presure (mmHg) | compare baseline data with 12 weeks rehabilitation data
depression scale by Patient Health Questionnaire | compare baseline data with 12 weeks rehabilitation data
  Patient Health Questionnaire (PHQ; range, 0-27; higher score = severe depression; cut-off score of 5 for minimal depression)
anxiety scale by Generalized Anxiety Disorder Scale | compare baseline data with 12 weeks rehabilitation data
  Generalized Anxiety Disorder Scale (GAD; range, 0-21; higher score = severe anxiety; cut-off score of 5 for mild anxiety)
fatigue scale by fatigue severity scale | compare baseline data with 12 weeks rehabilitation data
  fatigue severity scale (FSS; range, 9-63; higher score = severe fatigue; cut-off score of 4 for fatigue)
Quality of Life (QoL) questionnaire (MacNew) | compare baseline data with 12 weeks rehabilitation data
  MacNew QoL questionnaire is a measurement tool for patients with cardiac disease that measures physical, emotional, and social functional levels to provide overall QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Lim Joa, M.D., Principal Investigator — Department of physical medicine and rehabilitation, Inha University hospital
Locations (1):
- Inha University hospital, Incheon, Gyeonggi-do, South Korea